CLINICAL TRIAL: NCT03797703
Title: Efficacy of Lidocaine Gel Enema After Endoscopic Hemorrhoid Band Ligation for Relief of Post Procedural Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AHC-6999-M5000223
Record Dates: First submitted 2018-12-19; First posted 2019-01-09 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Patients will be randomly allocated into the treatment group. The treatment group will receive a 15 mL lidocaine gel enema rectally immediately following completion of the procedure.
  Interventions: Drug: Lidocaine Hydrochloride 2% gel enema
- Control (No Intervention): Patients will be randomly allocated into the control group. The control group will not receive a rectal enema.

INTERVENTIONS:
Drug: Lidocaine Hydrochloride 2% gel enema — Insertion of Lidocaine Hydrochloride 2% gel enema rectally immediately following the procedure.
  Arms: Treatment

SUMMARY:
This is a prospective study to assess the utility of Lidocaine Hydrochloride 2% gel enema (Hi-Tech Pharmacal Co., Inc.) in reducing post-procedural pain after endoscopic band ligation of internal hemorrhoids. Briefly, patients will be consented prior to entry into the study. During the endoscopic band ligation procedure, patients will be blindly placed into the treatment arm or control arm. The treatment arm will receive 15 ml enema of lidocaine gel immediately upon cessation of the procedure. In the placebo arm, oral pain medications will be provided. Researchers will assess pain following the procedure at 1 hour, 24 hours and 48 hours via telephone call. Another telephone call will be performed at 72 to 96 hours to assess any side effects of the medication.

DETAILED DESCRIPTION:
This is a prospective single center study to evaluate side effects and efficacy of a lidocaine jelly 2% enema following endoscopic hemorrhoid band ligation. The investigators will administer a single dose of 15 mL lidocaine jelly 2%, obtained from Advocate main pharmacy, as an enema immediately post procedure. Patients will not be permitted to self-administer additional doses following discharge.

Prior to being enrolled in the study, the clinician will perform a Comprehensive Metabolic Panel and Complete Blood Count. When appropriate, a urine pregnancy test will be performed prior to enrollment. The investigators will assess for any signs or symptoms of liver disease. These assessments will occur within one month of the procedure date. If the patient has any signs of renal or hepatic impairment (creatinine greater than 2 or Childs Pugh Class 3), they will be excluded from the study. The researchers will also exclude patients with any history of arrhythmias or who are currently on anti-arrhythmic medications. Once the patient is deemed safe to proceed, the lidocaine gel enema will be placed at the cessation of the procedure by the investigator. At the time of the procedure, the clinician will assess and use their best judgement to determine if the rectal mucosa is generally intact by visual inspection. If the mucosa remains intact, the subject will be able to be included in the study. However, if the rectal mucosa is traumatized the subject will be excluded and will not participate in the randomized treatment.

Following the procedure, the patient will be monitored closely with a one-on one registered nurse for 4 hours in an observation unit. Vital signs will be taken every 5 minutes, as well as continuous EKG monitoring and pulse oximetry monitoring. If any adverse side effects occur, the physician is immediately available for further management and admission to the hospital if needed. Upon completion of the 4-hour observation period, the participants will be evaluated by a registered nurse and physician prior to discharge home following the procedure. The patient will be discharged with a responsible adult who will care for the patient for 24 additional hours. The clinician will communicate with the patient and responsible adult regarding any adverse side effects. The patient will also receive a phone number to call to reach the physician or the physician's associate who will be able to verbally assist the patient immediately should any adverse events occur.

For data collection, one hour following the procedure a clinician will screen for any adverse side effects and pain will be assessed using a numeric pain scale (0-10). The patient will also be contacted via telephone to assess adverse side effects and pain scale at 24 hours and 48 hours post procedure. The investigators will also call the patient at 72 to 96 hours to assess for any adverse effects. The patients will be followed up by the principal investigator for routine check-ups following the procedure. The clinician will be easily accessible via telephone and the patient will be given instructions on how to contact the clinician, if needed.

Data to be collected on each subject will include: date of procedure, specific patient ID, gender, age, internal hemorrhoids grade, race (White, African American, Hispanic, Asian), BMI, comorbid conditions, pain 1 hour post procedure, pain 24 and 48 hours post procedure, requirement of narcotic pain medication, requirement of other oral analgesic medication, sedation utilized and complications or adverse side effects from the medication.

Upon data collection of this trial, we will monitor for any adverse events. If there is an adverse event that is deemed by the principal investigator likely due to drug administration, we will report it to the FDA immediately through written communication and an IND Safety Report. It will be reported within at least 7 calendar days of being notified of the adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* Patients undergoing endoscopic hemorrhoid band ligation at Advocate Christ Medical Center

Exclusion Criteria:

* Patients undergoing endoscopic hemorrhoids band ligation who are already on pain medications chronically due to other reasons
* Patients with moderate to severe renal impairment, defined as creatinine greater than 2
* Patients with hepatic dysfunction, defined as patients with signs or symptoms of liver dysfunction and/or patients with Childs Pugh Class C
* Patients with any history of arrhythmias or are currently on anti-arrhythmic medications
* Patients with any contraindications to lidocaine, including hypersensitivity to local anesthetics of the amide type or any other component within the lidocaine 2% jelly
* Patients with traumatized rectal mucosa in the area of application at the time of the procedure
* Patients who are currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Change in Pain following Procedure at 1 hour, 24 hours and 48 hours | This information will be collected at 1 hour, 24 hours and 48 hours after the procedure.
  This effect will be measured by statistical analysis comparing the treatment groups numeric pain scale ratings (0-10) with the control groups numeric pain scale ratings (0-10).

SECONDARY OUTCOMES:
Pain Medication Needs | This will be evaluated 48 hours after the procedure.
  This effect will be measured by asking the subject what pain medication was needed following the procedure and the amount taken.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Berkelhammer, MD, Principal Investigator — advocate christ medical center
Locations (1):
- Advocate Christ Medical Center, Oak Lawn, Illinois, United States

IPD SHARING:
Plan to Share IPD: No